CLINICAL TRIAL: NCT06318221
Title: A Randomized Clinical Trial With Perioperative Immunonutrition Support on Anthropometric, Clinical and Biochemical Parameters of Head and Neck Cancer Patients Undergoing Surgery
Brief Title: Effects of Perioperative Immunonutrition in Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Eda Başmısırlı, Asst. Prof. Dr., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06156930
Record Dates: First submitted 2024-02-15; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer; Nutrition, Healthy
Keywords: head and neck cancer; immunonutrition; enteral nutrition; Perioperative nutrition; Nutritional counseling
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Immunonutrition Diet; Population Groups

STUDY DESIGN:
Intervention Model Description: Patients were classified according to tumor location (oral cavity, oropharynx, larynx or hypopharynx) and body weight loss, approximately equally in both groups. Accordingly, patients were randomly assigned (by computer) into either the immunonutrition (intervention group) or standard EN (control group) groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immunonutrition (intervention group) (Experimental): Immunonutrition enteral products was given to the patients in the intervention group
  Interventions: Dietary Supplement: Experimental (Immunonutrition) Group
- standard (control group) (Active Comparator): Standard enteral products was given to patients in the control group.
  Interventions: Dietary Supplement: Active Comparator Group ( Standard enteral nutrition)

INTERVENTIONS:
Dietary Supplement: Experimental (Immunonutrition) Group — Immunonutrition was given to the patients in the intervention group and ready-to-use liquid in addition to their normal nutrition 5 days before the operation. The patients were instructed to consume three enteral products per day as taken between meals.
  In the postoperative period, feeding was started in the first 24 hours with the NG tube placed during the operation. The ready-to-use immunonutrition product was given to the patients in the intervention group.
  Arms: immunonutrition (intervention group)
Dietary Supplement: Active Comparator Group ( Standard enteral nutrition) — Standard enteral nutrition was given to patients in the control group in addition to their normal nutrition 5 days before the operation. The patients were instructed to consume three enteral products per day between meals.
  In the postoperative period, feeding was started in the first 24 hours with the NG tube placed during the operation. Liquid standard enteral nutrition was given to the patients in the control group.
  Arms: standard (control group)

SUMMARY:
A prospective randomized controlled study compared the effects of perioperative immunonutrition and standard enteral nutrition (EN) on postoperative short-term outcomes of patients with head and neck (HNC).

Five days before surgery and the postoperative day 10, immunonutrition support was given to the intervention group (n=17), and standard EN support was given to the control group (n=17). Body analyses were made, food consumption records were taken, NRS-2002 and quality of life scales were applied, and biochemical parameters were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx who will undergo surgery,
* who agree to receive standard EN or immunonutrition before surgery,
* those between the ages of 18-75,
* those with normal hematopoietic (absolute neutrophil count >1.8x109/L, hemoglobin level ≥9 g/dL) hepatic and renal function

Exclusion Criteria:

* Patients receiving neoadjuvant chemotherapy or radiotherapy to the head and neck region;
* Received EN support before the study
* have an active infection, any autoimmune, renal or hepatic disease, malabsorption, type 1 diabetes or mental illness
* taking vitamin-mineral supplements and immunosuppressive treatment,
* Morbidly obese (BMI ≥40 kg/m2), HIV positive, pregnant and breastfeeding individuals

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Body weight | 40 days
  Kg
Body weight loss | 40 days
  Kg
Body mass index | 40 days
  kg/m2
Resting metabolic rate | 40 days
  kcal
Nutrition Risk Screening 2002 | 40 days
  A total score of ≥3 indicates that the patient is at nutritional risk
The EORTC Core Quality of Life questionnaire-30 (EORTC QLQ-C30) | 40 days
  1. Estimate the average of the items that contribute to the scale; this is the raw score.
  2. Use a linear transformation to standardise the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
The EORTC Quality of life - Head and Neck Cancer Module (EORTC QLQ-H & N35) | 40 days
  The head & neck cancer module incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact and sexuality. There are also eleven single items. For all items and scales, high scores indicate more problems (i.e. there are no function scales in which high scores would mean better functioning).
Albumin | 40 days
  g/dL
C-reactive protein | 40 days
  mg/L
Prealbumin | 40 days
  mg/dL

SECONDARY OUTCOMES:
Length of hospital stay | 40 days
  days
Complication development status | 40 days
  It was evaluated as yes/no.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Talas, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No